CLINICAL TRIAL: NCT03267901
Title: Effects of Daily Walnut Intake Among the Subjects With Metabolic Syndrome in South Korea
Brief Title: Effects of Daily Walnut Intake Among the Subjects With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ICAN Nutrition Education and Research (Industry)
Collaborators: California Walnut Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CWC-2016-MetS
Record Dates: First submitted 2017-08-14; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Food

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walnut-Control (Experimental)
  Interventions: Other: food
- Control-Walnut (Experimental)
  Interventions: Other: food

INTERVENTIONS:
Other: food — 45 g of walnut / iso-caloric white bread

SUMMARY:
Investigators planed to conduct a randomized, controlled, crossover trial to examine the effects of daily walnuts intake among Korean subjects with metabolic syndrome. Primary objective of this study was to investigate the effects of daily walnut intake on changes of metabolic syndrome indices in Koreans with metabolic syndrome age over 30 years old. This study was consisted of four periods: run-in, first intervention, wash-out, and second intervention phases. As 16 weeks of first intervention period began after the run-in phase, the subjects were randomly assigned into one of two groups: walnut group and control group. Participants in walnut group consumed 45 grams of walnuts on a daily basis and participants in control group were provided iso-caloric white bread for first 16 weeks. After the first intervention and wash-out period (6 weeks), second intervention which is crossover of first intervention was started during the next 16 weeks. Anthropometric measurements and biochemical analyses were done at the beginning and the end of each intervention (0, 16, 22, and 38 weeks of trial). Habitual diet was randomly observed using 3-day diet record once during each phase.

Investigators expected to evaluate 1)effects of walnut ingestion on reverting metabolic syndrome to normal status especially by reducing waist circumference and improving serum levels of triglyceride and high-density lipoprotein, 2)beneficial effects of daily walnut consumption on changes of body composition in the subjects with metabolic syndrome, and 3)regulatory effects of daily walnut intake on inflammatory markers and diabetic markers.

ELIGIBILITY:
Inclusion Criteria: at least three out of five metabolic syndrome components

* waist circumference (WC) >90 cm for men and >80 cm for women
* hypertension (DBP ≥85 and <110 mm Hg)
* hyperglycemia (≥100 mg/dL)
* elevated plasma TG concentrations (≥150 mg/dL)
* decreased plasma HDL-C concentrations (<40 mg/dL for men and <50 mg/dL for women)

Exclusion Criteria:

* the presence of morbid obesity (BMI ≥40)
* the use of any medication for the control of blood pressure, glucose, or lipid metabolism
* a medical history of hypocaloric diet consumption within the past year
* gastrointestinal tract disorders
* post-menopausal women
* smokers

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
changes of waist circumference | after 16 weeks of daily walnut consumption
  Waist circumferences (cm) were obtained at the midpoint between the lowest rib and the iliac crest and rounded to the nearest 0.1 cm after inhalation and exhalation.
changes of blood triglyceride level | after 16 weeks of daily walnut consumption
  Serum triglycerides (mg/dL) levels were measured by an enzymatic-colorimetric method.
changes of blood high-density lipoprotein cholesterol levels | after 16 weeks of daily walnut consumption
  High density lipoprotein cholesterol (mg/dL) levels were determined by a homogeneous enzymatic-colorimetric method.
changes of blood pressure | after 16 weeks of daily walnut consumption
  Blood pressure (mmHg) was measured on the right arm using an up-load blood pressure monitor with participants in a comfortably seated position after at least a 5-minute rest.
changes of blood glucose level | after 16 weeks of daily walnut consumption
  Blood glucose levels (mg/dL) were measured using blood glucose monitor and test stripts from the finger tip.

SECONDARY OUTCOMES:
changes of total cholesterol level | after 16 weeks of daily walnut consumption
  Serum total cholesterol levels (ml/dL) were measured by an enzymatic-colorimetric method.
changes of serum apolipoprotein B level | after 16 weeks of daily walnut consumption
  Serum apolipoprotein B (ml/dL) was measured using a turbidimetric immunoassay.
changes of serum adiponectin level | after 16 weeks of daily walnut consumption
  Blood adiponectin (ug/mL) levels were measured using ELISA.
changes of serum leptin level | after 16 weeks of daily walnut consumption
  Blood leptin (ug/mL) levels were measured using ELISA.
changes of serum insulin level | after 16 weeks of daily walnut consumption
  Serum insulin (μU/mL) was measured with a commercially available kit, the ultrasensitive insulin ELISA kit using an Epoch microplate spectrophotometer.
changes of low-density lipoprotein cholesterol level | after 16 weeks of daily walnut consumption
  Low-density lipoprotein cholesterol levels (ml/dL) were determined by a homogeneous enzymatic-colorimetric method.

CONTACTS AND LOCATIONS:
Locations (1):
- ICAN Nutrition Education and Research, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hwang HJ, Liu Y, Kim HS, Lee H, Lim Y, Park H. Daily walnut intake improves metabolic syndrome status and increases circulating adiponectin levels: randomized controlled crossover trial. Nutr Res Pract. 2019 Apr;13(2):105-114. doi: 10.4162/nrp.2019.13.2.105. Epub 2019 Feb 11. PMID 30984354